CLINICAL TRIAL: NCT00806156
Title: A Multicenter, Open-Label, Phase 2 Study to Evaluate the Safety and Efficacy of NKTR-102 When Given on a Q14 Day or a Q21 Day Schedule in Patients With Metastatic or Locally Advanced Platinum-Resistant Ovarian Cancer
Brief Title: Study to Evaluate the Safety and Efficacy of NKTR-102 in Patients With Metastatic or Locally Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-PIR-04
Record Dates: First submitted 2008-12-04; First posted 2008-12-10 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Tumor; Ovarian Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NKTR-102 q14d (Experimental): NKTR-102 was administered as an intravenous (IV) infusion over 90 ± 10 minutes, on Day 1 of each 2-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 4 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Interventions: Drug: NKTR-102 q14d
- NKTR-102 q21d (Experimental): NKTR-102 was administered as an IV infusion over 90 ± 10 minutes, on Day 1 of each 3-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 6 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Interventions: Drug: NKTR-102 q21d

INTERVENTIONS:
Drug: NKTR-102 q14d — NKTR-102 given on a q14 day schedule
  Arms: NKTR-102 q14d
Drug: NKTR-102 q21d — NKTR-102 given on a q21 day schedule
  Arms: NKTR-102 q21d

SUMMARY:
This is a multicenter, open-label, two-arm, 2-stage, Phase 2 study of NKTR-102 in patients with metastatic or locally advanced platinum-resistant ovarian cancer.

Approximately 70 patients will be randomized 1:1 into one of two treatment arms. NKTR-102 will be administered at a dose level of 145 mg/m^2 in both arms. In Arm A, NKTR-102 will be given on a q14d schedule. In Arm B, NKTR-102 will be given on a q21d schedule. After the initial 70 patients have been enrolled, Arm B will enroll approximately 110 additional patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer
2. Inoperable metastatic or locally advanced ovarian cancer
3. Platinum-resistant ovarian cancer defined as progression by RECIST within 6 months of last dose of most recent platinum drug
4. Platinum-resistant patients who have progressed after receiving PLD (Doxil/Caelyx)therapy in a platinum-resistant setting or who otherwise unable to receive PLD therapy.
5. Diseases must be measurable as defined by RECIST in at least 1 lesion not previously irradiated.
6. ECOG performance score of 0 or 1.
7. Adequate organ and bone marrow functions at Screening.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) and have not recovered to NCI-CTCAE grade 1 toxicity prior to Day 1 of Cycle 1
2. Patients who have had any major surgery within 4 weeks prior to Day 1 of Cycle 1 or minor surgery within 2 weeks prior to Day 1 of Cycle 1
3. Patients who have received CYP3A4 inducers or inhibitors.
4. Patients who have received any treatment with a camptothecin derivative (eg. irinotecan, topotecan, SN38 investigational agents, etc.).
5. Patients with CNS metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (20):
- United States (11):
  - Investigator Site - Higland, Highland, California
  - Investigator Site - Los Angeles, Los Angeles, California
  - Investigator Site - Newport Beach, Newport Beach, California
  - Investigator Site - West Palm Beach, West Palm Beach, Florida
  - Investigator Site - Iowa City, Iowa City, Iowa
  - Investigator Site - Lansing, Lansing, Michigan
  - Investigator Site - Winston-Salem, Winston-Salem, North Carolina
  - Investigator Site - Oklahoma City, Oklahoma City, Oklahoma
  - Investigator Site - East Providence, East Providence, Rhode Island
  - Investigator Site - Nashville, Nashville, Tennessee
  - Investigator Site - Charlottesville, Charlottesville, Virginia
- Belgium (4):
  - Investigator Site - Gent, Ghent
  - Investigator Site - Leuven, Leuven
  - Investigator Site - Liege, Liège
  - Investigator Site - Wilrijk, Wilrijk
- United Kingdom (5):
  - Investigator Site - Middlesex, Middlesex, Northwood
  - Investigator Site - Coventry, Coventry
  - Investigator Site - Dundee, Dundee
  - Investigator Site - Glasgow, Glasgow
  - Investigator Site - Newcastle Upon Tyne, Newcastle upon Tyne

REFERENCES:
- [Derived] Rustin G, Vergote I, Micha JP, Duska LR, Reed N, Bendell J, Spitz D, Dark G, Hoch U, Tagliaferri M, Hannah AL, Garcia AA. A multicenter, open-label, expanded phase 2 study to evaluate the safety and efficacy of etirinotecan pegol, a polymer conjugate of irinotecan, in women with recurrent platinum-resistant or refractory ovarian cancer. Gynecol Oncol. 2017 Nov;147(2):276-282. doi: 10.1016/j.ygyno.2017.08.026. Epub 2017 Sep 19. PMID 28935273

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study began with an initial Simon two-stage design in which patients were randomized 1:1 into one of two treatment schedules (145 mg/m2 q14d or q21d). During Stage 1, 20 patients were to be enrolled and treated in each schedule (q14d or q21d). If at least 1 response was observed in 20 evaluable patients within a treatment schedule, the treatment schedule would progress to Stage 2, where an additional 15 patients were to be enrolled for a total of 35 patients in the treatment schedule.
Period: Overall Study
Arm/Group | NKTR-102 q14d | NKTR-102 q21d
Started | 39 | 139
Completed | 0 | 0
Not Completed | 39 | 139
Not completed — Death | 35 | 95
Not completed — Did not meet eligibility criteria | 1 | 0
Not completed — Study terminated by Sponsor | 2 | 40
Not completed — Consent withdrawn by subject | 1 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- NKTR-102 q14d: NKTR-102 was administered as an intravenous (IV) infusion over 90 ± 10 minutes, on Day 1 of each 2-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 4 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Note: NKTR-102 was administered at a dose level of 170 mg/m2 (10 patients enrolled and received this dose for 1 to 3 cycles) until the dose was reduced to 145 mg/m2 for all ongoing patients in the q14d and q21d treatment schedules and this became the starting dose for all newly enrolled patients. The dose was reduced based on safety results from ongoing NKTR-102 Phase 1 and 2 clinical studies and the reduction was initiated with a waiver for study sites.
- NKTR-102 q21d: NKTR-102 was administered as an IV infusion over 90 ± 10 minutes, on Day 1 of each 3-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 6 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Note: NKTR-102 was administered at a dose level of 170 mg/m2 (10 patients enrolled and received this dose for 1 to 3 cycles) until the dose was reduced to 145 mg/m2 for all ongoing patients in the q14d and q21d treatment schedules and this became the starting dose for all newly enrolled patients. The dose was reduced based on safety results from ongoing NKTR-102 Phase 1 and 2 clinical studies and the reduction was initiated with a waiver for study sites.
- Total: Total of all reporting groups
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Total
Number analyzed (Participants) | 39 | 139 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 99 | 126
  >=65 years | 12 | 40 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.14) | 58.3 (11.49) | 58.4 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 139 | 178
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST): Primary Efficacy Population
Description: The ORR was defined as the proportion of patients with a complete response (CR) or a partial response (PR) per RECIST 1.0 based upon the best response as assessed by the Investigator. CR was defined by RECIST 1.1 as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm. PR was defined by RECIST 1.1 as at least a 30% decrease in the sum of the diameters (SOD) of target lesions, taking as reference the baseline SOD. The analysis was performed for patients in the Primary Efficacy Population.
Time Frame: Every 6 weeks (± 5 days) from Cycle 1, Day 1 until documented disease progression, start of new therapy for cancer, death, or end of study (approximately 3 years and 11 months)
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- Primary Efficacy Population: The primary efficacy population consisted of patients in the modified intent-to-treat population (MITT) treated in q21d treatment schedule with platinum-resistant ovarian cancer who had received prior pegylated liposomal doxorubicin (PLD) therapy in a platinum-resistant setting or were otherwise unable to receive further PLD therapy.
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 104 | 104
Percentage of Patients | 14.4 [8.3 to 22.7] | 14.4 [8.3 to 22.7]

2. Secondary Outcome: Secondary: Best Overall Response by Gynecologic Cancer Intergroup (GCIG) Criteria: MITT Population
Description: Best overall response was defined as the proportion of patients with a CR or a PR as assessed per GCIG criteria. The GCIG proposed the following definition for the date of progression which used both the RECIST and cancer antigen 125 (CA-125) criteria. "A response according to CA-125 has occurred if there is ≥ 50% reduction in CA-125 levels from a pretreatment sample. The response had to be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA-125 only if they had a pretreatment sample that was at least twice the upper limit of normal (ULN) and within 2 weeks prior to starting treatment." Analysis was performed in MITT Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- NKTR-102 q14d; NKTR-102 q21d: NKTR-102 was administered as an IV infusion over 90 ± 10 minutes, on Day 1 of each 3-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 6 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Note: NKTR-102 was administered at a dose level of 170 mg/m2 (10 patients enrolled and received this dose for 1 to 3 cycles) until the dose was reduced to 145 mg/m2 for all ongoing patients in the q14d and q21d treatment schedules and this became the starting dose for all newly enrolled patients. The dose was reduced based on safety results from ongoing NKTR-102 Phase 1 and 2 clinical studies and the reduction was initiated with a waiver for study sites.
- MITT Population: The modified intent-to-treat (MITT) Population for the q14d Arm included all platinum-resistant ovarian cancer patients who were enrolled to the q14d treatment regimen. The MITT Population for the q21d Arm included all platinum-resistant ovarian cancer patients who were enrolled to the q21d treatment regimen. The MITT Population included those patients who had undergone radiographic tumor measurement evaluation at Baseline with measurable tumors, and were enrolled and received at least one dose (or partial dose) of study drug. Platinum-resistant patients had a platinum-free interval (PFI) ≤ 6 months. PFI was defined as the time to recurrence/progression from last dose of the prior platinum-based therapy.
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 37 | 132 | 169
Percentage of Patients | 29.7 [15.9 to 47] | 25 [17.9 to 33.3] | 26 [19.6 to 33.3]

3. Secondary Outcome: Secondary: Best Overall Response by GCIG Criteria: Primary Efficacy Population
Description: Best overall response was defined as the proportion of patients with a CR or a PR per assessed per GCIG criteria. The GCIG proposed the following definition for the date of progression which used both the RECIST and CA-125 criteria. "A response according to CA-125 has occurred if there is ≥ 50% reduction in CA-125 levels from a pretreatment sample. The response had to be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA-125 only if they had a pretreatment sample that was at least twice the ULN and within 2 weeks prior to starting treatment." Analysis was performed in Primary Efficacy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- Primary Efficacy Population: Patients in the MITT Population treated in q21d treatment schedule with platinum-resistant ovarian cancer, had received prior PLD therapy in a platinum-resistant setting or who were otherwise unable to receive further PLD therapy.
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 104 | 104
Percentage of Patients | 25 [17 to 34.4] | 25 [17 to 34.4]

4. Secondary Outcome: Secondary: Best Overall Response by GCIG Criteria: Platinum-Refractory Population
Description: Best overall response was defined as the proportion of patients with a CR or a PR per assessed per GCIG criteria. The GCIG proposed the following definition for the date of progression which used both the RECIST and CA-125 criteria. "A response according to CA-125 has occurred if there is ≥ 50% reduction in CA-125 levels from a pretreatment sample. The response had to be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA-125 only if they had a pretreatment sample that was at least twice the ULN and within 2 weeks prior to starting treatment." Analysis was performed in Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- Platinum-Refractory Population: Patients in the MITT Population with a PFI ≤ 6 weeks.
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 13 | 52 | 65
Percentage of Patients | 23.1 [5 to 53.8] | 17.3 [8.2 to 30.3] | 18.5 [9.9 to 30]

5. Secondary Outcome: Secondary: Best Overall Response by GCIG Criteria: Prior PLD Therapy Population
Description: Best overall response was defined as the proportion of patients with a CR or a PR per assessed per GCIG criteria. The GCIG proposed the following definition for the date of progression which used both the RECIST and CA-125 criteria. "A response according to CA-125 has occurred if there is ≥ 50% reduction in CA-125 levels from a pretreatment sample. The response had to be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA-125 only if they had a pretreatment sample that was at least twice the ULN and within 2 weeks prior to starting treatment." Analysis was performed in Prior PLD Therapy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- Prior PLD Population: Patients in the MITT Population treated in q14d and q21d treatment schedules, who subsequently progressed after receiving PLD therapy or who were otherwise unable to receive PLD therapy.
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 16 | 114 | 130
Percentage of Patients | 25 [7.3 to 52.4] | 24.6 [17 to 33.5] | 24.6 [17.5 to 32.9]

6. Secondary Outcome: Secondary: Kaplan-Meier Estimate of Progression-Free Survival (PFS): MITT Population
Description: According to enhanced RECIST 1.1, progressive disease was the appearance of one or more new lesions, OR an unambiguous increase in the sum of target lesion volumes with both 1) >20% increase in the sum of volumes (SOV) of all target lesions (taking as reference the nadir) and 2) greater than two times the variability of the measurements estimated by the sponsor and/or its designees.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 37 | 132 | 169
Months | 4.1 [2.6 to 6.7] | 4.4 [2.9 to 5] | 4.4 [3.1 to 5.3]

7. Secondary Outcome: Secondary: Kaplan-Meier Estimate of PFS: Primary Efficacy Population
Description: PFS was defined as the time from the date of the first NKTR-102 administration to the date of PD or death due to any cause. Progressive disease was determined by Investigators using RECIST criteria. Patients who were alive without disease progression at the time of data-cut-off were censored at the time of the last tumor assessment that demonstrated a lack of disease progression (or on Cycle 1 Day 1 if the patient did not undergo repeated imaging while on study). Analysis was performed in Primary Efficacy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 104 | 104
Months | 4.4 [2.9 to 5] | 4.4 [2.9 to 5]

8. Secondary Outcome: Secondary: Kaplan-Meier Estimate of PFS: Platinum-Refractory Population
Description: PFS was defined as the time from the date of the first NKTR-102 administration to the date of PD or death due to any cause. Progressive disease was determined by Investigators using RECIST criteria. Patients who were alive without disease progression at the time of data-cut-off were censored at the time of the last tumor assessment that demonstrated a lack of disease progression (or on Cycle 1 Day 1 if the patient did not undergo repeated imaging while on study). Analysis was performed in Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 13 | 52 | 65
Months | 11.9 [2 to 15] | 2.7 [1.7 to 4.6] | 3 [2 to 5.3]

9. Secondary Outcome: Secondary: Kaplan-Meier Estimate of PFS: Prior PLD Therapy Population
Description: PFS was defined as the time from the date of the first NKTR-102 administration to the date of PD or death due to any cause. Progressive disease was determined by Investigators using RECIST criteria. Patients who were alive without disease progression at the time of data-cut-off were censored at the time of the last tumor assessment that demonstrated a lack of disease progression (or on Cycle 1 Day 1 if the patient did not undergo repeated imaging while on study). Analysis was performed in Prior PLD Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 16 | 114 | 130
Months | 5.5 [2.2 to 11.4] | 4.4 [2.9 to 5] | 4.5 [3.1 to 5.3]

10. Secondary Outcome: Secondary: Kaplan-Meier Analysis of Duration of Overall Response (DoR): MITT Population
Description: DoR was defined as the time from the first documented CR or PR, the date of PD (assessed by central radiological review according to RECIST), or death due to any cause, whichever came first. Patients who were alive without documented PD per RECIST were censored at the date of last tumor assessment without disease progression or start of new anti-cancer therapy for the study disease, whichever was earlier. Analysis was performed in MITT Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 37 | 132 | 169
Months | 4.1 [2.8 to 8] | 6.6 [3.6 to 10.9] | 5.7 [4 to 10.1]

11. Secondary Outcome: Secondary: Kaplan-Meier Analysis of DoR: Primary Efficacy Population
Description: DoR was defined as the time from the first documented CR or PR, the date of PD (assessed by central radiological review according to RECIST), or death due to any cause, whichever came first. Patients who were alive without documented PD per RECIST were censored at the date of last tumor assessment without disease progression or start of new anti-cancer therapy for the study disease, whichever was earlier. Analysis was performed in Primary Efficacy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Primary Efficacy Population: The primary efficacy population consisted of patients with platinum-resistant ovarian cancer in the modified intent-to-treat population (MITT) treated in q21d treatment schedule who had received prior pegylated liposomal doxorubicin (PLD) therapy in a platinum-resistant setting or were otherwise unable to receive further PLD therapy.
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 104 | 104
Months | 7.4 [3.6 to 13.2] | 7.4 [3.6 to 13.2]

12. Secondary Outcome: Secondary: Kaplan-Meier Analysis of DoR: Platinum-Refractory Population
Description: DoR was defined as the time from the first documented CR or PR, the date of PD (assessed by central radiological review according to RECIST), or death due to any cause, whichever came first. Patients who were alive without documented PD per RECIST were censored at the date of last tumor assessment without disease progression or start of new anti-cancer therapy for the study disease, whichever was earlier. Analysis was performed in Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 13 | 52 | 65
Months | 10.8 [7.1 to 14.4] | 7.4 [2.9 to 12.6] | 7.4 [2.9 to 12.6]

13. Secondary Outcome: Secondary: Kaplan-Meier Analysis of DoR: Prior PLD Therapy Population
Description: DoR was defined as the time from the first documented CR or PR, the date of PD (assessed by central radiological review according to RECIST), or death due to any cause, whichever came first. Patients who were alive without documented PD per RECIST were censored at the date of last tumor assessment without disease progression or start of new anti-cancer therapy for the study disease, whichever was earlier. Analysis was performed in Prior PLD Therapy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 16 | 114 | 130
Months | 4.2 [4.1 to 14.4] | 7.4 [3.6 to 10.9] | 6.6 [4 to 10.9]

14. Secondary Outcome: Secondary: CA-125 Response Rate: MITT Population
Description: CA-125 response was determined by having achieved a ≥50% reduction in serum levels of CA-125 from a pre-treatment level of at least twice the ULN within 2 weeks of starting treatment according to the GCIG criteria. The CA-125 response rate was calculated as the number of patients meeting the endpoint definition divided by the total number of eligible patients per the GCIG criteria for CA-125 in the analysis population. Analysis was performed in MITT Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 32 | 109 | 141
Percentage of Patients | 43.8 [26.4 to 62.3] | 34.9 [26 to 44.6] | 36.9 [28.9 to 45.4]

15. Secondary Outcome: Secondary: CA-125 Response Rate: Primary Efficacy Population
Description: CA-125 response was determined by having achieved a ≥50% reduction in serum levels of CA-125 from a pre-treatment level of at least twice the ULN within 2 weeks of starting treatment according to the GCIG criteria. The CA-125 response rate was calculated as the number of patients meeting the endpoint definition divided by the total number of eligible patients per the GCIG criteria for CA-125 in the analysis population. Analysis was performed in Primary Efficacy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- Primary Efficacy Population: The primary efficacy population only included subjects treated in the NKTR-102 q21d treatment arm.
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 88 | 88
Percentage of Patients | 33 [23.3 to 43.8] | 33 [23.3 to 43.8]

16. Secondary Outcome: Secondary: CA-125 Response Rate: Platinum-Refractory Population
Description: CA-125 response was determined by having achieved a ≥50% reduction in serum levels of CA-125 from a pre-treatment level of at least twice the ULN within 2 weeks of starting treatment according to the GCIG criteria. The CA-125 response rate was calculated as the number of patients meeting the endpoint definition divided by the total number of eligible patients per the GCIG criteria for CA-125 in the analysis population. Analysis was performed in Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 11 | 40 | 51
Percentage of Patients | 36.4 [10.9 to 69.2] | 20 [9.1 to 35.6] | 23.5 [12.8 to 37.5]

17. Secondary Outcome: Secondary: CA-125 Response Rate: Prior PLD Therapy Population
Description: CA-125 response was determined by having achieved a ≥50% reduction in serum levels of CA-125 from a pre-treatment level of at least twice the ULN within 2 weeks of starting treatment according to the GCIG criteria. The CA-125 response rate was calculated as the number of patients meeting the endpoint definition divided by the total number of eligible patients per the GCIG criteria for CA-125 in the analysis population. Analysis was performed in Prior PLD Therapy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 15 | 95 | 110
Percentage of Patients | 40 [16.3 to 67.7] | 33.7 [24.3 to 44.1] | 34.5 [25.7 to 44.2]

18. Secondary Outcome: Secondary: Clinical Benefit Rate: MITT Population
Description: Clinical benefit rate was calculated as the number of patients with confirmed CR, PR, or SD (where the duration of SD should be ≥ 3 months) by RECIST divided by the total number of measurable patients in the population. Analysis was performed in MITT Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 37 | 132 | 169
Percentage of Patients | 56.8 [39.5 to 72.9] | 50.8 [41.9 to 59.6] | 52.1 [44.3 to 59.8]

19. Secondary Outcome: Secondary: Clinical Benefit Rate: Primary Efficacy Population
Description: Clinical benefit rate was calculated as the number of patients with confirmed CR, PR, or SD (where the duration of SD should be ≥ 3 months) by RECIST divided by the total number of measurable patients in the population. Analysis was performed in Primary Efficacy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 104 | 104
Percentage of Patients | 51 [41 to 60.9] | 51 [41 to 60.9]

20. Secondary Outcome: Secondary: Clinical Benefit Rate: Platinum-Refractory Population
Description: Clinical benefit rate was calculated as the number of patients with confirmed CR, PR, or SD (where the duration of SD should be ≥ 3 months) by RECIST divided by the total number of measurable patients in the population. Analysis was performed in Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 13 | 52 | 65
Percentage of Patients | 61.5 [31.6 to 86.1] | 38.5 [25.3 to 53] | 43.1 [30.8 to 56]

21. Secondary Outcome: Secondary: Clinical Benefit Rate: Prior PLD Therapy Population
Description: Clinical benefit rate was calculated as the number of patients with confirmed CR, PR, or SD (where the duration of SD should be ≥ 3 months) by RECIST divided by the total number of measurable patients in the population. Analysis was performed in Prior PLD Therapy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 16 | 114 | 130
Percentage of Patients | 56.3 [29.9 to 80.2] | 50.9 [41.3 to 60.4] | 51.5 [42.6 to 60.4]

22. Secondary Outcome: Secondary: Kaplan-Meier Analysis of Overall Survival (OS): MITT Population
Description: Duration of OS was defined as the time from the date of randomization to the date of death due to any cause. Patients were followed until their date of death, loss to follow-up, withdrawal of consent for further follow-up for survival, or final database closure. Patients who were lost-to-follow-up or were not known to have died were censored at last date they were shown to be alive. Patients who did not have any follow-up since the date of randomization were censored at the date of randomization. Analysis was performed in MITT Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 37 | 132 | 169
Months | 11.1 [8.8 to 16.7] | 10.2 [8.2 to 12.2] | 10.6 [9.4 to 12.2]

23. Secondary Outcome: Secondary: Kaplan-Meier Analysis of OS: Primary Efficacy Population
Description: Duration of OS was defined as the time from the date of randomization to the date of death due to any cause. Patients were followed until their date of death, loss to follow-up, withdrawal of consent for further follow-up for survival, or final database closure. Patients who were lost-to-follow-up or were not known to have died were censored at last date they were shown to be alive. Patients who did not have any follow-up since the date of randomization were censored at the date of randomization. Analysis was performed in Primary Efficacy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q21d | Primary Efficacy Population
Number analyzed (Participants) | 104 | 104
Months | 10.9 [8.2 to 13.1] | 10.9 [8.2 to 13.1]

24. Secondary Outcome: Secondary: Kaplan-Meier Analysis of OS: Platinum-Refractory Population
Description: Duration of OS was defined as the time from the date of randomization to the date of death due to any cause. Patients were followed until their date of death, loss to follow-up, withdrawal of consent for further follow-up for survival, or final database closure. Patients who were lost-to-follow-up or were not known to have died were censored at last date they were shown to be alive. Patients who did not have any follow-up since the date of randomization were censored at the date of randomization. Analysis was performed in Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 13 | 52 | 65
Months | 11.1 [6.1 to 21.6] | 8 [5 to 12.2] | 9.4 [5.8 to 12.2]

25. Secondary Outcome: Secondary: Kaplan-Meier Analysis of OS: Prior PLD Therapy Population
Description: Duration of OS was defined as the time from the date of randomization to the date of death due to any cause. Patients were followed until their date of death, loss to follow-up, withdrawal of consent for further follow-up for survival, or final database closure. Patients who were lost-to-follow-up or were not known to have died were censored at last date they were shown to be alive. Patients who did not have any follow-up since the date of randomization were censored at the date of randomization. Analysis was performed in Prior PLD Therapy Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 16 | 114 | 130
Months | 12.2 [8.8 to 16.7] | 11 [8.9 to 13.1] | 11 [9.5 to 12.5]

26. Secondary Outcome: Secondary: ORR by RECIST: MITT Population
Description: The ORR was defined as the proportion of patients with a CR or a PR per RECIST 1.0 based upon the best response as assessed by the Investigator assessment. The analysis was performed for patients in the MITT Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | MITT Population
Number analyzed (Participants) | 37 | 132 | 169
Percentage of Patients | 21.6 [9.8 to 38.2] | 15.2 [9.5 to 22.4] | 16.6 [11.3 to 23]

27. Secondary Outcome: Secondary: ORR by RECIST: Prior PLD Population
Description: The ORR was defined as the proportion of patients with a CR or a PR per RECIST 1.0 based upon the best response as assessed by the Investigator assessment. The analysis was performed for patients in the PLD Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Prior PLD Population
Number analyzed (Participants) | 16 | 114 | 130
Percentage of Patients | 18.8 [4 to 45.6] | 14.9 [8.9 to 22.8] | 15.4 [9.7 to 22.8]

28. Secondary Outcome: Secondary: ORR by RECIST: Platinum-Refractory Population
Description: The ORR was defined as the proportion of patients with a CR or a PR per RECIST 1.0 based upon the best response as assessed by the Investigator assessment. The analysis was performed for patients in the Platinum-Refractory Population.
Time Frame: as for outcome 1
Population: Received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- NKTR-102 q14d: NKTR-102 was administered as an intravenous (IV) infusion over 90 ± 10 minutes, on Day 1 of each 2-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 4 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Note: NKTR-102 was administered at a dose level of 170 mg/m2 (10 patients enrolled and received this dose for 1 to 3 cycles) until the dose was reduced to 145 mg/m2 for all ongoing patients in the q14d and q21d treatment schedules and this became the starting dose for all newly enrolled patients. The dose was reduced based on safety results from ongoing NKTR-102 Phase 1 and 2 clinical studies and the reduction was initiated with a waiver for study sites and shortly thereafter included in Protocol Amendment 1.0 dated 26 Mar 2009.
- NKTR-102 q21d: NKTR-102 was administered as an IV infusion over 90 ± 10 minutes, on Day 1 of each 3-week [± 2 days] cycle at a dose of 170 mg/m^2 for the first 6 patients enrolled and at a dose of 145 mg/m^2 for the remainder of the patients.
  Note: NKTR-102 was administered at a dose level of 170 mg/m2 (10 patients enrolled and received this dose for 1 to 3 cycles) until the dose was reduced to 145 mg/m2 for all ongoing patients in the q14d and q21d treatment schedules and this became the starting dose for all newly enrolled patients. The dose was reduced based on safety results from ongoing NKTR-102 Phase 1 and 2 clinical studies and the reduction was initiated with a waiver for study sites and shortly thereafter included in Protocol Amendment 1.0 dated 26 Mar 2009.
Arm/Group | NKTR-102 q14d | NKTR-102 q21d | Platinum-Refractory Population
Number analyzed (Participants) | 13 | 52 | 65
Percentage of Patients | 15.4 [1.9 to 45.4] | 15.4 [6.9 to 28.1] | 15.4 [7.6 to 26.5]

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study (approximately 3 years and 11 months).
Description: Safety Population=177 patients (n=38 NKTR-102 dose every 14 days; n=139 NKTR-102 dose every 21 days). All 177 participants experienced at least one adverse event, and 101 of them experienced at least one serious adverse event. Other Adverse Events section lists events occurring > 5% of patients.
Arm/Group | NKTR-102 q14d | NKTR-102 q21d
All-Cause Mortality (participants affected / at risk) | 35/38 | 95/139
Serious Adverse Events (participants affected / at risk) | 23/38 | 78/139
Other Adverse Events (participants affected / at risk) | 38/38 | 139/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-102 q14d (N=38) | NKTR-102 q21d (N=139)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 2 (2) | 11 (11)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombocytopenia subjects affected / (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cholinergic syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 7 (8)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (3)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 21 (24)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 7 (7)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (8)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 11 (19)
Vomiting (Gastrointestinal disorders) | 3 (3) | 9 (10)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 13 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 2 (2)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2)
Herpes oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-102 q14d (N=38) | NKTR-102 q21d (N=139)
Flushing (Vascular disorders) | 1 (3) | 9 (13)
Hypotension (Vascular disorders) | 3 (4) | 6 (6)
Asthenia (General disorders) | 3 (5) | 12 (16)
Chills (General disorders) | 2 (2) | 7 (11)
Fatigue (General disorders) | 20 (38) | 81 (198)
Oedema peripheral (General disorders) | 7 (10) | 15 (20)
Pyrexia (General disorders) | 11 (15) | 23 (33)
Anxiety (Psychiatric disorders) | 7 (8) | 12 (12)
Depression (Psychiatric disorders) | 3 (3) | 11 (13)
Insomnia (Psychiatric disorders) | 7 (8) | 15 (20)
Blood creatinine increased (Investigations) | 3 (3) | 10 (14)
Haemoglobin decreased (Investigations) | 1 (1) | 8 (16)
Weight decreased (Investigations) | 18 (31) | 42 (51)
Tachycardia (Cardiac disorders) | 2 (3) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 10 (19) | 38 (65)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 13 (43)
Neutropenia (Blood and lymphatic system disorders) | 9 (22) | 27 (74)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 8 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 13 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 28 (39)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
Dizziness (Nervous system disorders) | 11 (17) | 25 (36)
Dysgeusia (Nervous system disorders) | 8 (8) | 17 (24)
Headache (Nervous system disorders) | 6 (13) | 23 (42)
Lethargy (Nervous system disorders) | 2 (6) | 8 (13)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 6 (8)
Vision blurred (Eye disorders) | 9 (14) | 26 (41)
Abdominal distension (Gastrointestinal disorders) | 7 (8) | 17 (19)
Abdominal pain (Gastrointestinal disorders) | 16 (21) | 74 (128)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 10 (11)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 15 (22)
Ascites (Gastrointestinal disorders) | 3 (3) | 8 (12)
Constipation (Gastrointestinal disorders) | 9 (12) | 51 (87)
Diarrhoea (Gastrointestinal disorders) | 34 (230) | 103 (376)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 8 (14) | 17 (30)
Flatulence (Gastrointestinal disorders) | 8 (10) | 16 (19)
Nausea (Gastrointestinal disorders) | 27 (70) | 107 (250)
Stomatitis (Gastrointestinal disorders) | 3 (8) | 17 (20)
Vomiting (Gastrointestinal disorders) | 23 (54) | 76 (176)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (16) | 29 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 11 (12)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 17 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 15 (16)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 16 (25)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (13)
Decreased appetite (Metabolism and nutrition disorders) | 20 (35) | 69 (135)
Dehydration (Metabolism and nutrition disorders) | 11 (20) | 22 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (5) | 7 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (24) | 28 (61)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 8 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6) | 15 (28)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 7 (8)
Urinary tract infection (Infections and infestations) | 6 (7) | 11 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.